CLINICAL TRIAL: NCT03992989
Title: Quality Control of CE-Certified Phonak Hearing Aids - 2019_19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Sonova2019_19
Record Dates: First submitted 2019-06-19; First posted 2019-06-20 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Hearing Loss; Sensorineural Hearing Loss
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Sensorineural

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phonak Bolero M90-M (Experimental): The Phonak Bolero M90-M is a Behind-the-Ear Hearing aid with direct connectivity functionality from Phonak which will be fitted to the participants individual Hearing loss
  Interventions: Device: Phonak Bolero M90-M
- Roger Select (Active Comparator): The Roger Select is an accessory which can be connected to a compatible hearing aid. It offers an external microphone which streams signals directly to the connected hearing aid.
  Interventions: Device: Roger Select

INTERVENTIONS:
Device: Phonak Bolero M90-M — The Phonak Bolero M90-M is a Behind-the-Ear Hearing aid with direct connectivity functionality from Phonak which will be fitted to the participants individual Hearing loss
  Arms: Phonak Bolero M90-M
Device: Roger Select — The Roger Select is an accessory which can be connected to a compatible hearing aid. It offers an external microphone which streams signals directly to the connected hearing aid.
  Arms: Roger Select

SUMMARY:
Phonak Hearing Systems pass through different development and study stages. At an early stage, feasibility studies are conducted to investigate new algorithms, features and functions in an isolated manner. If the benefit is proven, their performance is then investigated regarding interdependency between all available algorithms, features and functions running in parallel in a hearing aid (pivotal/pre-validation studies) and, as a result, they get optimized. Afterwards, and prior to product launch, the Phonak Hearing Systems undergo a final quality control in terms of clinical trials. This is a pre-validation study, investigating optimized algorithms, features, functions and wearing comfort. This will be a clinical evaluation which will be conducted mono centric at Sonova AG Headquarters based in Stäfa (Switzerland).

DETAILED DESCRIPTION:
In this study one CE-labeled Phonak Behind-the-ear (BTE) devices is investigated including CE-labeled compatible accessories. The experimental device will be investigated regarding its performance of speech understanding in noise with and without an accessory existing of an external microphone to pick sound at a certain target. A secondary objective of this study is the investigation of the Overall system stability in daily life situations. The experimental device contains direct connectivity functionality. Another objective of this study is the investigation of the subjective occlusion effect of different acoustic couplings. This will be a clinical evaluation which will be conducted mono centric at Sonova AG Headquarters based in Stäfa (Switzerland).

ELIGIBILITY:
Inclusion Criteria:

* Adult hearing impaired persons (minimum age: 18 years, mild to moderate Hearing loss) without hearing aid experience
* Good written and spoken (Swiss) German language skills
* Healthy outer ear
* Ability to fill in a questionnaire (p/eCRF) conscientiously
* Informed Consent as documented by signature
* owning a compatible smartphone
* Hearing loss in range of N2-N3 (ISO 60118-15)

Exclusion Criteria:

* Contraindications to the MD in this study, e.g. known hypersensitivity or allergy to the investigational product
* Limited mobility and not in the position to attend weekly appointments in Stäfa (Switzerland)
* Limited ability to describe listening impressions/experiences and the use of the hearing aid
* Inability to produce a reliable hearing test result
* Known psychological problems
* Central hearing disorders

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2019-07-06 (Actual); Study Completion 2019-07-06 (Actual)

PRIMARY OUTCOMES:
Speech intelligibility in noise | 1 week
  The primary objective of this study is to investigate the speech intelligibility in noise of the investigational device alone versus the active comparator. Speech understanding in noise will be evaluated with an objective and validated test procedure, the Outcome measure will be the value of speech intelligibility in percentage at a certain signal to noise ratio.

SECONDARY OUTCOMES:
Subjective Sound quality perception | 4 weeks
  The secondary objective of this study is to investigate the overall sound quality perception of the investigational device for daily real life situations. The sound quality perception will be measured with a subjective satisfaction rating scale ranging from 0% to 100%.

OTHER OUTCOMES:
Subjective occlusion effect | 4 weeks
  Another objective of this study is to investigate the subjectively perceived occlusion effect of the own voice by the use of the investigational device. The subjective occlusion effect will be investigated with subjective ratings scales for the dimensions 'dullness of own voice' and 'naturalness of own voice'
Sound quality for streamed audio signals | 1 week
  Another objective of this study is to evaluate the subjectively perceived sound quality of streamed audio signals [via bluetooth streaming] with the help of a subjective rating scale

CONTACTS AND LOCATIONS:
Locations (1):
- Sonova AG, Stäfa, Canton of Zurich, Switzerland